CLINICAL TRIAL: NCT00577577
Title: A Placebo Controlled, Randomized, Double-Blind Phase II Clinical Trial to Evaluate Tolerability, Safety and Efficacy Endpoints After Administration of Recombinant Human Insulin-Like Growth Factor-I/Recombinant Human Insulin-Like Growth Factor Binding Protein-3 (rhIGF-I/rhIGFBP-3) for 24 Weeks in Adults With Myotonic Dystrophy Type 1
Brief Title: Safety and Efficacy Study of Recombinant Human Insulin-Like Growth Factor-I/Recombinant Human Insulin-Like Growth Factor Binding Protein-3 (rhIGF-I/rhIGFBP-3) In Myotonic Dystrophy Type 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: INSM-110-1001
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Myotonic Dystrophy Type 1
MeSH Terms: conditions — Myotonic Dystrophy | interventions — Insulin-Like Growth Factor I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhIGF-I/rhIGFBP-3 (Experimental)
  Interventions: Drug: rhIGF-I/rhIGFBP-3
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rhIGF-I/rhIGFBP-3 — 1.0 mg/kg rhIGF-I/rhIGFBP-3 or placebo daily, subcutaneous injections from baseline through the last day of the end of study visit.
  Arms: rhIGF-I/rhIGFBP-3
Drug: placebo — 1.0 mg/kg rhIGF-I/rhIGFBP-3 or placebo daily, subcutaneous injections from baseline through the last day of the end of study visit.
  Arms: Placebo

SUMMARY:
To investigate the effects of rhIGF-I/rhIGFBP-3 treatment for 24 weeks on endurance, ambulation, cognitive functioning, insulin resistance, lipid levels, muscle function and strength, pain, gastrointestinal functioning, and quality of life endpoints in DM1 patients

DETAILED DESCRIPTION:
Efficacy Measures:

Endurance, Ambulation, Cognitive function, Insulin resistance, Cholesterol and triglycerides, Muscle function and strength, Pain, Gastrointestinal function, Quality of life

MINIMUM INCLUSION CRITERIA

1. A diagnosis of DM1, confirmed by DM1 genetic mutation
2. Age 21 to 65 years (inclusive)
3. Ability to walk 30 feet - assistance with cane and/or leg bracing permitted
4. Able to self-administer study medication by subcutaneous injection or caregiver is available to administer study medication

ELIGIBILITY:
Inclusion Criteria (list is not inclusive):

* A diagnosis of DM1, confirmed by DM1 genetic mutation
* Ability to walk 30 feet - assistance with cane and/or leg bracing permitted
* Able to self-administer study medication by subcutaneous injection or caregiver is available to administer study medication

Exclusion Criteria (list is not inclusive):

* Congenital DM1
* Weight greater than 100 kg or body mass index greater than 30 kg/m2
* Prior treatment with glucocorticoids, anabolic steroids, testosterone, growth hormone, investigational agent within 60 days of screening
* Current diagnosis or history of malignancy expect for surgically cured skin cancer or pilomatricoma
* Changes in lipid lowering medications during the 3 months prior to screening
* Diaphragmatic weakness such that patients are unable to tolerate the supine position, or swallowing impairment such that patients are unable to maintain nutrition without use of gastrostomy.
* Major psychiatric illness (major depression, bipolar disorder or schizophrenia) within twelve months of screening
* History of non-compliance with other therapies

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2008-12-29 (Actual); Study Completion 2008-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Moxley, M.D., Study Chair — University of Rochester Neuromuscular Disease Center
Locations (12):
- United States (12):
  - University of California Irvine Medical Center; MDA, ALS and Neuromuscular Center, Orange, California
  - University of California, Davis, Sacramento, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - University of Rochester, Neuromuscular Disease Center, Rochester, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregan Health and Science University, Portland, Oregon
  - Universit of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 13 research centers in the United States from December 2007 to December 2008.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either IPLEX™ (Recombinant Human Insulin-Like Growth Factor-I/Recombinant Human Insulin-Like Growth Factor Binding Protein-3 [rhIGF-I/rhIGFBP-3]) or matched placebo for 24 weeks.
Groups:
- IPLEX™: Participants received 1.0 mg/kg IPLEX™ (rhIGF-I/rhIGFBP-3) via a subcutaneous injection once a day for 24 weeks.
- Placebo: Participants received a matching placebo to IPLEX™ once a day via a subcutaneous injection for 24 weeks.
Period: Overall Study
Arm/Group | IPLEX™ | Placebo
Started | 34 | 35
Received Treatment | 34 | 35
Completed | 29 | 30
Not Completed | 5 | 5
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 3
Not completed — Transportation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) population: all enrolled participants who had at least one dose of IPLEX™ or placebo and had at least one post-baseline efficacy assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | IPLEX™ | Placebo | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 35 | 69
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.36 (8.74) | 44.17 (10.40) | 45.25 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 18 | 16 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not collected. Population: Ethnicity was not collected.
  Participants
    Hispanic or Latino | 1 | 2 | 3
    Not Hispanic or Latino | 33 | 33 | 66
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 30 | 33 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Distance Walked as Assessed by the Six-minute Walk Test (6MWT) Distance
Description: The 6MWT measured the distance in meters that participants were able to walk over a total of six minutes. After a 10 minute resting period, the participants completed the 6MWT on a hard, flat surface at baseline and at Week 24.
Time Frame: Baseline and Week 24
Population: Per protocol (PP) population: all enrolled participants who were at least 80% compliant with study dosing, had no more than 21 days interruption in therapy at any one time, had efficacy assessments required at the Week 24 study visit, met all inclusion and exclusion criteria, and were not major protocol violators. Only participants with data available for analysis are reported.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 25 | 27
meters | 12.40 (44.75) | 20.11 (50.87)

2. Primary Outcome: Change From Baseline in Daily Step Count
Description: The number of steps taken per day was measured using a step activity monitor for 7 days at baseline and again at Week 24. Change from baseline scores were measured where a negative change from baseline indicates a decrease in the number of daily steps.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: daily step count
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 13 | 20
daily step count | -140 (1222) | -58 (1209)

3. Primary Outcome: Peak Activity Index: Change From Baseline in Number of Steps Walked Per Minute During the 30 Minute Period of Fastest Walking
Description: The peak activity index measures the number of steps walked in the 30 minutes of fastest walking that occurred in a 24 hour period. This was measured using a step activity monitor for 7 days at baseline and again at Week 24. Change from baseline scores were measured where a positive change from baseline indicates an improvement in the number of steps walked during the 30 minute period of fastest walking.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steps per minute (steps/min)
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 13 | 20
steps per minute (steps/min) | 0.5 (6.9) | 1.1 (6.0)

4. Primary Outcome: Sustained Activity Index: Change From Baseline in the Highest Number of Steps Walked Per Minute Over 20 Minutes of Activity
Description: The sustained activity index measures the highest number of steps sustained over a continuous 20 minute period. This was measured using a step activity monitor for 7 days at baseline and again at Week 24. Change from baseline scores were measured where a positive change from baseline indicates an improvement in the number of steps walked over 20 minutes of activity.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steps per minute (steps/min)
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 13 | 20
steps per minute (steps/min) | -0.9 (8.3) | 0.8 (5.9)

5. Primary Outcome: Change From Baseline in the Percentage of Time That Participants Spent Inactive
Description: Change from baseline scores were measured where a negative change from baseline indicates less time spent inactive.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 13 | 20
percentage of time | -0.4 (6.6) | -0.0 (5.2)

6. Primary Outcome: Change From Baseline in Time Taken for Participants to Ascend and Descend 4 Stairs
Description: Participants were timed on their ability to climb up 4 stairs and timed separately to climb down 4 stairs at baseline and at week 24. The stairs were free-standing or the same flight of stairs was used at each assessment. Change from baseline scores were measured where a positive change from baseline indicates an improvement in the time taken for paticipants to ascend or descend 4 stairs.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 23 | 25
seconds
  Ascend 4 stairs | 0.0 (0.8) | -0.5 (1.2)
  Descend 4 stairs: number analyzed (Participants) | 22 | 25
  Descend 4 stairs | -0.1 (1.0) | -0.5 (1.5)

7. Primary Outcome: Change From Baseline in Time Taken to Traverse 30 Feet
Description: Participants were timed on their ability to travel 30 feet on the same surface at each assessment at baseline and at Week 24. Change from baseline scores were measured where a positive change from baseline indicates an improvement in the time taken to travel 30 feet.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 24 | 27
seconds | 0.2 (1.3) | -0.2 (2.2)

8. Primary Outcome: Change From Baseline in Purdue Pegboard Test Scores
Description: The Purdue Pegboard Test consists of a board with two sets of 25 holes, 4 concave cups, and a number of small metal pins. Participants were required to pick up the pins from a holder and place them in the holes as quickly as possible over 30 seconds with their dominant hand. The score was calculated as the number of pins placed into holes in 30 seconds and was measured at baseline and Week 24. Change from baseline scores were measured where a positive change from baseline indicates an improvement in the number of pins placed in the board.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of pins
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 25 | 29
number of pins | -0.2 (2.4) | 0.3 (1.5)

9. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Volume While Sitting or Lying Down
Description: FVC is the volume of air that can be forcibly exhaled from the lungs after taking the deepest breath possible, as measured by spirometry.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 23 | 28
litres
  Sitting FVC | -0.1 (0.3) | 0.0 (0.5)
  Lying down FVC: number analyzed (Participants) | 22 | 26
  Lying down FVC | -0.2 (0.4) | -0.1 (0.3)

10. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Percent Predicted While Sitting or Lying Down
Description: as for outcome 9
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage (%) of FVC predicted
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 22 | 27
Percentage (%) of FVC predicted
  Sitting FVC (%) | 0.0 (6.8) | -2.3 (11.0)
  Lying Down FVC (%): number analyzed (Participants) | 22 | 25
  Lying Down FVC (%) | -3.8 (8.4) | -3.2 (11.1)

11. Primary Outcome: Change From Baseline in Manual Muscle Test (MMT) Scores
Description: The MMT was used to assess muscle strength in the distal muscles and the proximal muscles. Distal muscles assessments included wrist extension, wrist flexion, ankle dorsiflexion and plantarflexion. Proximal muscle assessments included shoulder abduction, elbow extension, elbow flexion, hip extension, hip abduction, hip flexion, knee extension and knee flexion.
  In MMT, each muscle assessment was given a score of 0 to 5, where 0 indicated 'no contraction palpable' and 5 indicated 'normal strength'. The scores from each muscle were summed and the maximum overall score of all measured muscles was 140, the maximum distal score was 40 and the maximum proximal score was 80. Higher scores indicated higher muscle strength. Change from baseline scores were measured where a positive change from baseline indicates an improvement in muscle strength.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 24 | 29
Score on a scale
  Overall Score: number analyzed (Participants) | 23 | 27
  Overall Score | 0.9 (7.0) | -0.3 (4.0)
  Distal Muscles: number analyzed (Participants) | 24 | 28
  Distal Muscles | -0.4 (3.0) | 0.0 (1.5)
  Proximal Muscles: number analyzed (Participants) | 23 | 29
  Proximal Muscles | 1.0 (4.4) | -0.3 (2.9)

12. Primary Outcome: Change From Baseline in Selective Reminding Test T-Scores (Total Word and Delayed Words)
Description: The Selective Reminding Test measures verbal learning and memory and involves remembering a verbal list of 12 words. Participants were required to recall the 12 words presented. Words that were missed on recall were presented again, and the process was repeated until all 12 words were correctly recalled. The total word list recall and delayed recall were calculated as T-scores. Raw scores were converted to T-score using available normative data. Change from baseline T-scores were measured where a positive change from baseline indicates improvement in performance.
Time Frame: Baseline and Week 24
Population: Modified Per Protocol Population:
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 21 | 25
T-score
  Word List T-Score | 4.3 (7.4) | 2.9 (8.9)
  Delayed Recall T-Score | -3.2 (8.2) | 0.04 (7.8)

13. Primary Outcome: Change From Baseline in Selective Reminding Test Raw Scores (Cued Recall and Recognition)
Description: The Selective Reminding Test measures verbal learning and memory and involves remembering a verbal list of 12 words. Participants were required to recall the 12 words presented. Words that were missed on recall were presented again, and the process is repeated until all 12 words were correctly recalled. The cued recall scores ranged from 0-11 and multiple choice recognition scores ranged from 0-12. Change from baseline scores were measured where a positive change from baseline indicates an improvement in verbal recall and memory.
Time Frame: Baseline and Week 24
Population: Modified Per Protocol Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 21 | 25
Score on a scale
  Cued Recall Raw Score | 0.0 (0.9) | -0.4 (0.9)
  Recognition Raw Score | 0.0 (0.4) | 0 (0.4)

14. Primary Outcome: Change From Baseline in Rey Complex Figure (RCF) Test Scores
Description: The Rey Complex Figure Test (RCFT) assesses visuospatial construction ability and visual memory through four different tests: copy (copying a complex geometric figure), immediate recall of the figure (drawing figure from memory at 3 minutes), delayed recall (drawing figure at 30 minutes after initial copy), and recognition score (selecting individual parts of the figure from sketches provided). Copy performances are divided into 18 components with a maximum score of 2 each. The maximum score for each figure is 36.
Time Frame: Baseline and Week 24
Population: Modified Per Protocol Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 22 | 27
Score on a scale
  Immediate Recall T-Score | 7.5 (7.9) | 4.8 (11.4)
  Delayed Recall T-Score: number analyzed (Participants) | 22 | 25
  Delayed Recall T-Score | 5.2 (8.5) | 4.8 (11.7)
  Recognition T-Score: number analyzed (Participants) | 22 | 26
  Recognition T-Score | -1.5 (14.3) | 5.9 (12.7)

15. Primary Outcome: Change From Baseline in Letter-Number Sequencing (LNS) Test Scores
Description: The LNS test from the Welchsler Adult Intelligence Scale-III was used to assess working memory. The test required that participants recall, in order, numbers and letters presented in an unordered sequence. The number of items is 21. With each item being marked 0 if reported incorrectly or 1 if reported correctly, the maximum score is 21. Raw scores were converted into T-scores using available normative data. Change from baseline T-scores were measured where a positive change from baseline indicates improvement in performance.
Time Frame: Baseline and Week 24
Population: Intention to treat (ITT) population: all enrolled participants who had at least one dose of IPLEX™ or placebo and had at least one post-baseline efficacy assessment. Only participants with data available for analysis are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 28 | 33
Score on a scale | 1.18 (3.64) | -0.36 (2.09)

16. Primary Outcome: Change From Baseline in Trail Making Test (TMT) Scores
Description: The TMT assesses executive function, sequencing, mental flexibility, visual spanning speed and motor function. In TMT Part A, the participant had to draw lines in the correct order between 25 numbers randomly arranged on the page. In TMT Part B, the participant had to draw lines between 25 numbers and letters in alternating order (e.g., 1-A-2-B...etc). Times for Part A and Part B were used to derive T-scores which can range from a minimum of 0 and a maximum of 100. Raw scores were converted into T-scores using available normative data. Change from baseline T-scores were measured where a positive change from baseline indicates improvement in performance.
Time Frame: Baseline and Week 24
Population: Modified Per Protocol Population
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 22 | 27
T-score
  TMT Part A | 2.2 (10.2) | -0.3 (9.1)
  TMT Part B | 4.0 (7.1) | -0.9 (8.9)

17. Primary Outcome: Change From Baseline in the Stroop Color Word Test Scores
Description: The Stroop Color Word Test measures selective attention and cognitive flexibility. The test has three parts, the Word test (reading words), the Color test (naming the ink color in which words are displayed) and the Color-Word test (saying the ink color not reading the word). An interference score was calculated from the Color, Word and Color-Word scores and is an indication of how well a person can complete a task while disregarding interfering information. Raw scores were converted into T-scores using available normative data. Scores range from 0 to 100. Change from baseline T-scores were measured where a positive change from baseline indicates improvement in performance.
Time Frame: Baseline and Week 24
Population: Modified Per Protocol Population
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 22 | 25
T-score
  Word T-Score | -0.4 (7.0) | 2.0 (6.8)
  Color T-Score: number analyzed (Participants) | 22 | 24
  Color T-Score | 2.0 (4.1) | 0.9 (5.5)
  Color-Word T-Score: number analyzed (Participants) | 21 | 23
  Color-Word T-Score | 1.3 (4.6) | 1.0 (7.3)
  Interference T-Score: number analyzed (Participants) | 21 | 23
  Interference T-Score | 0.9 (4.6) | -0.2 (7.5)

18. Primary Outcome: Change From Baseline to Week 24 Scores on the Beck Depression Inventory II (BDI-II) Questionnaire
Description: BDI-II is a validated self-reported instrument of 21 questions which are each scored 0-3. Total scores range from 0-63, with higher score totals indicating more severe depression symptoms. {0-9: indicates minimal depression; 0-18: indicates mild depression; 19-29: indicates moderate depression; 30-63: indicates severe depression. Lower scores indicate no or minimal depression, with a maximum total score of 63.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 24 | 28
Score on a scale | -1.63 (6.34) | -0.14 (5.44)

19. Primary Outcome: Change From Baseline in Average Fasting Glucose Concentration in the Blood
Description: Participants were administered 75 grams (g) glucose solution prior to administration of the first dose of IPlex™ and after administration of the last dose. A 2-hour oral glucose tolerance test (OGTT) was performed under fasted conditions.
Time Frame: Baseline - Pre-dose and 30, 60, 90 and 120 minutes post glucose solution; Week 24 - Pre-dose and 30, 60, 90 and 120 minutes post glucose solution
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 21 | 25
milligrams per deciliter (mg/dL) | -6.8 (9.5) | 0.2 (10.5)

20. Primary Outcome: Change From Baseline in Average Fasting Insulin Concentration in the Blood
Description: Participants were administered 75 g glucose solution prior to administration of the first dose of IPLEX™ and after administration of the last dose. A 2-hour OGTT was performed under fasted conditions.
Time Frame: as for outcome 19
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: micro units per milliliter (μU/mL)
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 21 | 25
micro units per milliliter (μU/mL) | -5.7 (7.7) | 0.7 (8.8)

21. Primary Outcome: Change From Baseline in Qualitative Insulin Sensitivity Check Index (QUICKI)
Description: The QUICKI is based on fasting glucose and insulin measurements and are calculated using the following equation:
  QUICKI = 1/[ log(fasting glucose in mg/dL) + log (fasting insulin in uU/mL) ]
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 21 | 25
Index | 0.05 (0.04) | -0.01 (0.05)

22. Primary Outcome: Change From Baseline in Insulin Sensitivity Index-Matsuda (ISI-Matsuda)
Description: The ISI-Matsuda is based on the average glucose and insulin values obtained during the entire oral glucose tolerance test and are calculated using the following equation:
  ISI = 10,000 / √ [ fasting glucose (mg/dL) x fasting insulin(uU/mL) x mean glucose x mean insulin ]
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 17 | 23
Index | 5.5 (3.2) | -1.4 (3.6)

23. Primary Outcome: Change From Baseline in Total Blood Cholesterol Level
Description: A negative change from baseline indicates a decrease in total blood cholesterol level.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 25 | 26
mg/dL | -7.9 (20.4) | -2.7 (30.1)

24. Primary Outcome: Change From Baseline in Total Blood Low-density Lipoproteins (LDL) Level
Description: A positive change from baseline indicates an increase in total blood LDL level.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams per milliliter (mg/mL)
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 24 | 23
milligrams per milliliter (mg/mL) | 1.5 (18.2) | 5.0 (20.9)

25. Primary Outcome: Change From Baseline in Total Blood High-density Lipoproteins (HDL) Level
Description: A negative change from baseline indicates a decrease in total blood HDL level.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 25 | 26
mg/dL | 0.3 (9.9) | -3.0 (7.5)

26. Primary Outcome: Change From Baseline in Total Blood Triglycerides Level
Description: A negative change from baseline indicates a decrease in total blood triglycerides level.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 25 | 26
mg/mL | -54.8 (87.6) | -21.7 (105.9)

27. Primary Outcome: Change From Baseline in Gastro-esophageal Reflux Disease (GERD) Symptom Frequency Questionnaire (GSFQ) Scores
Description: The GSFQ contains 6 questions that assess the frequency of certain GERD symptoms and their impact on daily life. Scores were converted and reported out of 100 with higher scores indicative of more frequent and intense GERD symptoms. Change from baseline scores were measured where a negative change from baseline indicates less frequent and intense GERD symptoms.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 25 | 29
Score on a scale | -6.4 (11.8) | -0.5 (8.8)

28. Primary Outcome: Change From Baseline in Gastrointestinal Symptom Rating Scale for Irritable Bowel Syndrome (GSRS-IBS) Questionnaire Scores
Description: The GSRS-IBS has 13 questions aimed at identifying the frequency and intensity of IBS symptoms during the past week. Answers are given a score from 1 (no discomfort at all) to 7 (very severe discomfort). A total score was calculated and ranged from 0 to 78. A lower score indicates less discomfort from IBS symptoms. Change from baseline scores were measured where a positive change from baseline indicates increased discomfort from IBS symptoms.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 25 | 29
Score on a scale | -0.29 (0.63) | -0.02 (0.83)

29. Primary Outcome: Change From Baseline in Swallowing Disturbance Questionnaire (SDQ) Scores
Description: The SDQ had 15 questions relating to the oral phase and pharyngeal phase of swallowing. Answers for 14 questions were assigned a number (0-3) based on a 4-point verbal scale (never, seldom, frequently, very frequently) and the last question was a yes or no question about respiratory infections. A higher score is indicative of greater swallowing issues with 44.5 as the highest possible score. A total score of ≥ 11 suggests impairment. Change from baseline scores were measured where a positive change from baseline indicates increased swallowing impairment.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 24 | 29
Score on a scale | 0.29 (3.3) | -0.34 (4.4)

30. Primary Outcome: Change From Baseline in Short Form (36) (SF-36) Questionnaire Scores
Description: The SF-36 is a 36-item questionnaire that evaluates quality of life through physical and mental health across eight scales, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability. Change from baseline scores were measured where a positive change from baseline indicates an improvement in quality of life.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 25 | 29
Score on a scale
  Physical Health | 1.4 (6.9) | -0.5 (5.7)
  Mental Health | 1.2 (7.3) | 1.2 (9.1)

31. Primary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Questionnaire - Severity Scores
Description: The BPI contains 15 questions that assess the severity of pain and its impact or interference on functions of daily life. Pain severity was measured as the mean of 7 items of the questionnaire on an 11-point scale where 0 indicates no pain and 10 indicates the worst pain. A higher score indicates greater pain. Categories assessed include worst pain in 24 hours and average pain. Change from baseline scores were measured where a positive change from baseline indicates a worsening in pain.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 25 | 29
Score on a scale
  Worst pain in 24 hours | 0.0 (2.6) | 0.5 (2.7)
  Average pain | -0.2 (2.4) | 0.6 (2.1)

32. Primary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Questionnaire - Interference Scores
Description: The BPI contains 15 questions that assess the severity of pain and its impact or interference on functions of daily life. Pain interference is measured as the mean of 7 items on an 11-point scale where 0 indicates no interference and 10 indicates complete interference. A higher score indicates greater impairment due to pain. Change from baseline scores were measured where a positive change from baseline indicates a worsening of interference due to pain.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | IPLEX™ | Placebo
Number analyzed (Participants) | 23 | 26
Score on a scale | 0.0 (1.6) | -0.5 (1.6)

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: All-cause mortality and serious adverse events are reported for all participants enrolled/randomized in the study. Other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | IPLEX™ | Placebo
All-Cause Mortality (participants affected / at risk) | 1/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 7/34 | 6/35
Other Adverse Events (participants affected / at risk) | 31/34 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPLEX™ (N=34) | Placebo (N=35)
Bundle Branch Block Left (Cardiac disorders) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Chest Pain (Cardiac disorders) | 0 | 1
Ventricular Dysfunction (Cardiac disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Headache (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPLEX™ (N=34) | Placebo (N=35)
Ear Pain (Ear and labyrinth disorders) | 2 | 0
Vision Blurred (Eye disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Consitpation (Gastrointestinal disorders) | 8 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 3
Stomach Discomfort (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 2 | 1
Fatigue (General disorders) | 4 | 5
Injection Site Bruising (General disorders) | 3 | 8
Hyperhidrosis (General disorders) | 2 | 1
Oedema (General disorders) | 2 | 0
Oedema Peripheral (General disorders) | 5 | 2
Pyrexia (General disorders) | 2 | 1
Influenza (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 3
Urinary Tract Infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 5
Joint Sprain (Injury, poisoning and procedural complications) | 3 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Balance Disorder (Nervous system disorders) | 2 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 9 | 3
Hypoaethesia (Nervous system disorders) | 3 | 2
Insomnia (Nervous system disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 2 | 1
Depression (Psychiatric disorders) | 2 | 2
Irritability (Psychiatric disorders) | 2 | 0
Endometriosis (Reproductive system and breast disorders) | 2 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Rash Papular (Skin and subcutaneous tissue disorders) | 2 | 1
Injection Site Burning (General disorders) | 0 | 4
Injection Site Erythema (General disorders) | 12 | 3
Injection Site Haemorrhage (General disorders) | 1 | 2
Injection Site Pain (General disorders) | 11 | 7
Injection Site Pruritus (General disorders) | 7 | 0
Injection Site Swelling (General disorders) | 2 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Chest Pain (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0
Epidermal Naevus (Congenital, familial and genetic disorders) | 1 | 0
Ear Disorder (Ear and labyrinth disorders) | 1 | 0
Ear Infection (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Corneal Abrasion (Eye disorders) | 1 | 0
Eye Swelling (Eye disorders) | 0 | 1
Retinal Haemorrhage (Eye disorders) | 0 | 1
Visual Field Defect (Eye disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Change of Bowel Habit (Gastrointestinal disorders) | 1 | 0
Defaecation Urgency (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastroenteritis Viral (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Energy Increased (General disorders) | 1 | 1
Gait Abnormal (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1
Injection Site Induration (General disorders) | 1 | 0
Injection Site Urticaria (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Rigors (General disorders) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Eye and Eyelid Infections (Infections and infestations) | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 6
Back Injury (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1
Mouth Injury (Injury, poisoning and procedural complications) | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Ejection Fraction Decreased (Investigations) | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1
High Density Lipoprotein Decreased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0
Oestradiol Increased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0
Transaminases Increased (Investigations) | 0 | 1
Weight Increased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Increased Appetite (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw Inflammation (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 1
Burning Sensation (Nervous system disorders) | 1 | 0
Disturbance in Attention (Nervous system disorders) | 1 | 0
Dysphonia (Nervous system disorders) | 0 | 1
Hyporeflexia (Nervous system disorders) | 1 | 0
Sensory Loss (Nervous system disorders) | 1 | 0
Sinus Headache (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Panic Disorder (Psychiatric disorders) | 1 | 0
Staring (Psychiatric disorders) | 1 | 0
Stress Symptoms (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Batholin's Cyst (Reproductive system and breast disorders) | 0 | 1
Breast Tenderness (Reproductive system and breast disorders) | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea Exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Periorbital Haematoma (Vascular disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No